CLINICAL TRIAL: NCT06983275
Title: Exploration of the Effectiveness of Vibrational Intervention in Improving Insomnia Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jia Xiu (Other)
Collaborators: Shanghai Minhang Central Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Nanjing Brain Hospital affiliated with Nanjing Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Jia Xiu, doctoral student, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vibrational sleep intervention
Record Dates: First submitted 2025-05-10; First posted 2025-05-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia; vibrational neuromodulation; vibration
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The control group is designed to serve as a comparison to the intervention group, to determine whether the intervention produces real therapeutic effects. Participants in the control group will take part in a 9-week study, consisting of:
  1. Week 1 (Adaptation Phase): Daily sleep diary recording
  2. Weeks 2-5 (Intervention Phase): Daily sham stimulation and sleep diary recording
  3. Weeks 6-9 (Follow-up Phase): Daily sleep diary recording Memory performance assessments will be conducted within one week following the adaptation phase and again within one week after the follow-up phase. Participants will also complete a sleep questionnaire once per week throughout the study.
  Interventions: Other: Sham
- Intervention group (Experimental): The intervention group is designed to verify whether the stimulation yields true therapeutic effects in comparison to the control group. Participants in the intervention group will also undergo a 9-week study, consisting of:
  1. Week 1 (Adaptation Phase): Daily sleep diary recording
  2. Weeks 2-5 (Intervention Phase): Daily active stimulation and sleep diary recording
  3. Weeks 6-9 (Follow-up Phase): Daily sleep diary recording Memory performance assessments will be conducted within one week following the adaptation phase and again within one week after the follow-up phase. Participants will complete a sleep questionnaire once per week throughout the study.
  Interventions: Device: Vibrational stimulation

INTERVENTIONS:
Device: Vibrational stimulation — Fifteen minutes before bedtime, participants will wear a vibration stimulation device on the forehead while lying down in a comfortable position. The stimulation intensity will be set to 60% of the device's maximum output. Participants will receive a 15-minute session of 40 Hz vibration stimulation with a 50% duty cycle: 15 seconds of stimulation followed by 15 seconds of rest, repeated continuously. After the session, participants will remove the device and prepare for sleep immediately.
  Arms: Intervention group
Other: Sham — Fifteen minutes before bedtime, participants will lie down in a comfortable position and listen to the 40 Hz noise generated by the vibration device (without receiving actual vibration). After the session, they will remove the device and prepare for sleep immediately.
  Arms: Control group

SUMMARY:
Study Purpose The purpose of this clinical trial is to investigate whether low-intensity frontal vibration can improve sleep performance in individuals with chronic insomnia. Additionally, the study aims to explore its potential effects on memory enhancement.

The primary objectives of the study are to address the following questions:

* Does low-intensity frontal vibration improve sleep performance in patients with chronic insomnia?
* Does low-intensity frontal vibration enhance memory performance in patients with chronic insomnia?

Researchers will compare the effects of low-intensity frontal vibration with a sham stimulation (in which participants hear only noise associated with the vibration process) to determine whether the active intervention can effectively improve symptoms of chronic insomnia.

Participant Involvement

Participants in the study will:

* Record daily sleep diaries via a mobile application for a total of 9 weeks
* Receive daily intervention during a 4-week intervention phase as scheduled by the study
* Complete weekly self-reported sleep questionnaires through the app
* Undergo memory performance assessments at the beginning and end of the study

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years, regardless of gender;
* Diagnosed with chronic insomnia disorder according to DSM-5 criteria, with a primary complaint of difficulty falling asleep (sleep onset latency > 30 minutes), occurring ≥3 times per week, lasting for more than 3 months but less than 3 years;
* Able to independently operate a smartphone, and capable of completing self-reported assessments and applying the self-administered intervention after instruction.

Exclusion Criteria:

* Presence of sleep disorders such as sleep apnea syndrome or restless legs syndrome;
* Epworth Sleepiness Scale (ESS) score > 10;
* Use of any sleep-related medication within the past month;
* Patient Health Questionnaire-9 (PHQ-9) score > 15 or Generalized Anxiety Disorder-7 (GAD-7) score > 10;
* Currently participating in any form of cognitive behavioral therapy or neuromodulation intervention study;
* Working night shifts or rotating shifts;
* Clinically diagnosed neurological disorders such as epilepsy, stroke, dementia, or Parkinson's disease, or psychiatric disorders such as bipolar disorder, obsessive-compulsive disorder, phobias, or panic disorder;
* Substance abuse (including alcohol or drugs), defined as more than 14 drinks/week for males or 12 drinks/week for females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index Scale(PSQI) | baseline(Day 1); intervention stage(The last day of each week during 4-week intervention); follow-up stage(The last day of each week during 4-week follow-up)
  A scale that evaluates sleep quality, the scale scores range from 0 to 21, and lower scores mean a better outcome

SECONDARY OUTCOMES:
The Insomnia Severity Index Scale(ISI) | baseline(Day 1); intervention stage(The last day of each week during 4-week intervention); follow-up stage(The last day of each weekduring 4-week follow-up)
  A scale that evaluates the severity of insomnia, the scale scores range from 0 to 28, and lower scores mean a better outcome
Epworth Sleepiness Scale(ESS) | baseline(Day 1); intervention stage(The last day of each week during 4-week intervention); follow-up stage(The last day of each week during 4-week follow-up)
  A scale that evaluates sleepiness, the scale scores range from 0 to 24, and lower scores mean a better outcome
Patient Health Questionnaire (PHQ-9) | baseline(Day 1); intervention stage(The last day of each week during 4-week intervention); follow-up stage(The last day of each week during 4-week follow-up)
  A scale that evaluates the severity of depression, the scale scores range from 0 to 27, and lower scores mean a better outcome
Generalized Anxiety Disorder-7 (GAD-7) | baseline(Day 1); intervention stage(The last day of each week during 4-week intervention); follow-up stage(The last day of each week during 4-week follow-up)
  A scale that evaluates anxiety, the scale scores range from 0 to 21, and lower scores mean a better outcome
Sleep Diary | Daily recording for the duration of the 63-day trial.
  A sleep diary is a record of an individual's sleep and wake times, also sleep performence.
Memory Task | baseline(Day 1); intervention stage(The last day of 4-week intervention, an average of Day 35); follow-up stage(The last day 4-week stage, an average of Day 63)
  This task involves the sequential presentation of 40 pairs of nouns on a screen. Each word pair is displayed for 4 seconds, with a 1-second interval between pairs. The words within each pair are semantically related (e.g., brain - consciousness).
  Following the learning phase, participants complete an immediate cued-recall test. During this test, the first word of each pair is presented in a randomized order, and the participant is asked to verbally recall the second word. There is no time limit for each response. After each attempt, the correct answer is immediately displayed on the screen as feedback.
  Approximately 30 minutes later, a delayed recall test is administered using the same cued-recall procedure. However, no feedback is provided after the responses during this delayed test.
  Recall performance from both time points is used to calculate the offline gain in memory performance, defined as:
  Offline Gain (%) = ((Post-sleep Recall / Pre-sleep Rec
Intervention Experience | through study completion, an average of 63 days
  Participants will be asked whether they experienced any discomfort during the intervention and to rate the perceived effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Refer the information in publication